CLINICAL TRIAL: NCT06659614
Title: Prostate Tissue Biobank for People at Genetic Risk for Aggressive Disease
Brief Title: Prostate Tissue BioBank
Acronym: PTBB
Status: Recruiting | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Principal Investigator, Kara Maxwell, Principal investigator, Abramson Cancer Center at Penn Medicine
Other Study IDs: UPCC 21823; IRB 854327 (Other: University of Pennsylvania)
Record Dates: First submitted 2024-10-24; First posted 2024-10-26 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Prostate Cancer; Genetic Predisposition
MeSH Terms: conditions — Prostatic Neoplasms; Genetic Predisposition to Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Collecting biospecimens including blood and tissue. DNA may be derived from either sample type. Tissue biospecimens will be collected from primary prostate biopsy via needle core biopsy, prostatectomy and metastatic soft tissue and bone biopsy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Carriers: Eligible subjects will have confirmed pathogenic or likely pathogenic variants in a prostate cancer risk gene, and will also be undergoing prostate needle biopsy, prostatectomy or metastatic biopsy. Study participation will request access to medical information, blood and tissue samples.
- Controls: Eligible subjects will be undergoing prostate needle biopsy, prostatectomy or metastatic biopsy. Study participation will request access to medical information, blood and tissue samples.

SUMMARY:
Prostate cancer is also the most common cancer in men with inherited pathogenic variants in BRCA1 and BRCA2. Beyond BRCA1/2, other genes are known to increase the risk of prostate cancer, including ATM, TP53 and HOXB13. The investigators have shown that 5% of men diagnosed with prostate cancer localized to their prostate gland and up to 10-15% of patients with metastatic prostate cancer gland are carriers of an inherited gene mutation.

The Prostate Tissue BioBank is a prospective study which aims to create a biorepository of prostate tissue samples from prostate biopsies and prostatectomies and matched germline DNA from pathogenic mutation carriers in addition to age-matched control samples. Our primary goal is to investigate prostate cancer development and treatment response in carriers of germline DNA repair mutations, as compared to non-carrier controls.

ELIGIBILITY:
Inclusion Criteria:

Carriers (Group 1):

1. Confirmed pathogenic or likely pathogenic variant in a known prostate cancer risk gene.
2. Patients undergoing prostate biopsies as a part of their prostate cancer screening OR biopsy or prostatectomy due to a diagnosis of prostate cancer

Controls (Group 2):

1. Patients undergoing prostate biopsies as a part of their prostate cancer screening OR biopsy or prostatectomy due to a diagnosis of prostate cancer

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People assigned male at birth, undergoing prostate biopsies as a part of their prostate cancer screening OR biopsy or prostatectomy due to a diagnosis of prostate cancer
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2034-01 (Estimated); Study Completion 2034-01 (Estimated)

PRIMARY OUTCOMES:
Clinical and pathological data for patients with prostate tissue samples | 5 years
  Data will be collected on consented patients who undergo prostate biopsy, prostatectomy or metastatic biopsy.

CONTACTS AND LOCATIONS:
Overall Officials: Kara N Maxwell, MD, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided
Study participant research data will be securely stored by the study investigators. Any plan to share this data will require a Data Use Agreement executed and approved by the University of Pennsylvania.